CLINICAL TRIAL: NCT06002568
Title: ) The Effect of Intraoperative Binaural Beats on the Quantity of Inhaled Anesthetic Gas Required for the Maintenance of General Anesthesia: a Randomized, Placebo Controlled Trial
Brief Title: Effect of Binaural Beats for Maintenance of General Anesthesia
Acronym: BB
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 2306-028-1437
Record Dates: First submitted 2023-07-25; First posted 2023-08-21 (Actual); Last update posted 2023-08-21 (Actual); Status verified 2023-07

CONDITIONS: Anesthesia, General
Keywords: Sevoflurane; Brain waves; Binaural Beats

STUDY DESIGN:
Intervention Model Description: A prospective randomized, placebo-controlled trial
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (Placebo Comparator): In the control group, a silent state (a wave file made without sound) is applied via the sound generator and a headset, at the starting of general anesthesia induction. The sound generator volume is set to 60 dB. The sound generator and the headset is assigned after the randomization, and is blinded to the patient and the investigator. This sound is applied during the operation, and at the time of the final skin suture, the sound generator and the headset will be removed from the patient.
  Interventions: Procedure: Silent
- Binaural Beat (Experimental): In the experimental group, the binaural beat which is produced by the beat of 1Hz difference is applied via the sound generator and a headset, at the starting of general anesthesia induction. The sound generator volume is set to 60 dB. The sound generator and the headset is assigned after the randomization, and is blinded to the patient and the investigator. This sound is applied during the operation, and at the time of the final skin suture, the sound generator and the headset will be removed from the patient.
  Interventions: Procedure: Binaural beats

INTERVENTIONS:
Procedure: Silent — Apply wave file created in silence.
  Arms: Control
Procedure: Binaural beats — Apply wave file which is intended to generate binaural beats by applying waves of different frequency (1Hz difference) in each ear.
  Arms: Binaural Beat

SUMMARY:
The goal of this clinical trial is to learn about the effects of binaural beats on maintenance of general anesthesia in patients undergoing thyroidectomy without intraoperative neuromonitoring.

The main question it aims to answer is:

* 1) Does applying binaural beats during surgery reduce the gas anesthetics (especially sevoflurane) requirement to maintaining adequate anesthetic depth during general anesthesia?
* 2) Does applying binaural beats during surgery affect intraoperative hemodynamic stability or post operative nausea and vomiting?

Participants will wear headsets with a sound generator which contains music files (binaural beat file in the intervention group (BB) ; silent file in control group (C)) according to the randomization. Researchers will compare the BB and C group to see if intraoperative binaural beats reduce the requirements of sevoflurane for maintaining adequate anesthetic depth.

DETAILED DESCRIPTION:
This study will look at thyroidectomy patients without neuromonitoring. Before entering the operating room, patients will be randomized according to the randomization table, with the test group receiving a sound generating device with a binaural sound file and the control group receiving a sound generating device with a silent file. After entering the operating room, electrocardiogram, pulse oxymetry, non-invasive blood pressure monitor, and sensor for depth of anesthesia will be attached. At the beginning of anesthesia induction, the headset will be placed on the patient and a sound generator will be connected to the headset to play the file. The induction of anesthesia will be done with administration of fentanyl and propofol in both groups, and after confirming that the patient is unresponsive to voice, rocuronium and sevoflurane will be administrated to the patient. During the operation, the inhaled anesthetic concentration will be adjusted to maintain a patient state index (PSI) between 25 and 50. Fentanyl can be titrated up to 100 mcg to account for the hemodynamic response to intraoperative pain, and neuromuscular blocking agents are titrated to maintain a train of four (TOF) count of 1-3. The headset is continuously applied to the patient during surgery, and blood pressure, pulse oximetry, PSI, end tidal sevoflurane and end tidal minimal alveolar concentration will be monitored during the operation. At the time of the final suture of the skin, the sound generator will be removed from the headset. Save the raw EEG data from the Sedline® sensor for further analytical evaluation.

ELIGIBILITY:
Inclusion Criteria:

* Patients who are scheduled for thyroidectomy without neuromonitoring
* Patients aged 20-60 who require general anesthesia over 2 hours
* Patients who are able to provide written consent to participate in the clinical trial, to understand the procedure of this clinical trial, and to fill out the questionnaire appropriately
* Patients with ASA physical status classification 1-2

Exclusion Criteria:

* Patients with hearing loss or using hearing aids
* Patients who received narcotic analgesics or sedative drugs within 1 week
* Patients with alcohol or drug dependence
* Patients with drug hypersensitivity to sevoflurane
* Patients with family history or past history of malignant hyperthermia
* Patients with neuromuscular disease of myasthenia gravis
* Patients with arrhythmia, cardiovascular disease, and decreased heart function
* Patients with kidney failure
* Patients who are judged to be inappropriate for this clinical trial according to the opinions of investigators

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 122 (Estimated)
Dates: Start 2023-08 (Estimated); Primary Completion 2025-07-29 (Estimated); Study Completion 2025-07-31 (Estimated)

PRIMARY OUTCOMES:
Average end tidal sevoflurane concentration | From the starting of surgery to the final suture of skin
  Average end tidal sevoflurane concentrations required for maintenance of general anesthesia from surgical incision to skin closure

SECONDARY OUTCOMES:
End tidal minimal alveolar concentration - Maximum | From the starting of surgery to the final suture of skin
  Maximal value of end tidal minimal alveolar concentration during maintenance of general anesthesia
End tidal minimal alveolar concentration - Minimum | From the starting of surgery to the final suture of skin
  Minimal value of end tidal minimal alveolar concentration during maintenance of general anesthesia
Anxiety | Right after arriving the operating room
  Anxiety is evaluated using visual analogue score(0-100mm ruler without a scale), after entering the operating room
Anxiety | Just before leaving the post anesthesia care unit
  Anxiety is evaluated using visual analogue score(0-100mm ruler without a scale), just before leaving the post anesthesia care unit
Vital sign | From the starting to the end of general anesthesia
  Noninvasive blood pressure (systolic & diastolic & mean, mmHg)
Vital sign | From the starting to the end of general anesthesia
  Heart rate (bpm)
Vital sign | From the starting to the end of general anesthesia
  Saturation by pulse oximeter (%)
Brain wave | From the starting of surgery to the final suture of skin
  Patient state index (PSI) by Sedline device
Brain wave | From the starting of surgery to the final suture of skin
  brainwaves (raw data) which are collected in the Sedline device - alpha, beta, theta, delta, gamma brain wave
Post operative nausea vomiting | During the patients stay in post anesthesia care unit
  The incidence of post operative nausea vomiting, in the post anesthesia care unit
Post operative nausea vomiting | Since the patient leaves the post anesthesia care unit, until post operative 24 hours
  The incidence of post operative nausea vomiting, in the ward within 24 hours
Post operative pain | While the patient stay in post anesthesia care unit
  Pain is evaluate in Numerical rating scales score (0-10, 0 for no pain and 10 for for worst pain imaginable), in the post anesthesia care unit
Post operative pain | 24 hours after operation
  Pain is evaluate in Numerical rating scales score (0-10, 0 for no pain and 10 for for worst pain imaginable), 24 hours after operation
Delirium | Since the patient leaves the post anesthesia care unit, until post operative 24 hours
  The incidence of delirium in the ward within 24 hours after operation
Delirium | Since the patient leaves the post anesthesia care unit, until post operative 48 hours
  The incidence of delirium in the ward within 48 hours after operation

CONTACTS AND LOCATIONS:
Overall Officials: Jeong-Hwa Seo, MD., PhD., Principal Investigator — Seoul National University Hospital
Locations (1):
- Seoul National University Hospital, Seoul, South Korea

REFERENCES:
- [Background] American Society of Anesthesiologists Task Force on Intraoperative Awareness. Practice advisory for intraoperative awareness and brain function monitoring: a report by the american society of anesthesiologists task force on intraoperative awareness. Anesthesiology. 2006 Apr;104(4):847-64. doi: 10.1097/00000542-200604000-00031. No abstract available. PMID 16571982
- [Background] Torri G. Inhalation anesthetics: a review. Minerva Anestesiol. 2010 Mar;76(3):215-28. PMID 20203550
- [Background] Saller T, Hubig L, Seibold H, Schroeder Z, Wang B, Groene P, Perneczky R, von Dossow V, Hinske LC. Association between post-operative delirium and use of volatile anesthetics in the elderly: A real-world big data approach. J Clin Anesth. 2022 Dec;83:110957. doi: 10.1016/j.jclinane.2022.110957. Epub 2022 Sep 6. PMID 36084424
- [Background] Vutskits L, Xie Z. Lasting impact of general anaesthesia on the brain: mechanisms and relevance. Nat Rev Neurosci. 2016 Oct 18;17(11):705-717. doi: 10.1038/nrn.2016.128. PMID 27752068
- [Background] Ji D, Karlik J. Neurotoxic Impact of Individual Anesthetic Agents on the Developing Brain. Children (Basel). 2022 Nov 19;9(11):1779. doi: 10.3390/children9111779. PMID 36421228
- [Background] Wilder RT, Flick RP, Sprung J, Katusic SK, Barbaresi WJ, Mickelson C, Gleich SJ, Schroeder DR, Weaver AL, Warner DO. Early exposure to anesthesia and learning disabilities in a population-based birth cohort. Anesthesiology. 2009 Apr;110(4):796-804. doi: 10.1097/01.anes.0000344728.34332.5d. PMID 19293700
- [Background] Block RI, Thomas JJ, Bayman EO, Choi JY, Kimble KK, Todd MM. Are anesthesia and surgery during infancy associated with altered academic performance during childhood? Anesthesiology. 2012 Sep;117(3):494-503. doi: 10.1097/ALN.0b013e3182644684. PMID 22801049
- [Background] Fu VX, Sleurink KJ, Janssen JC, Wijnhoven BPL, Jeekel J, Klimek M. Perception of auditory stimuli during general anesthesia and its effects on patient outcomes: a systematic review and meta-analysis. Can J Anaesth. 2021 Aug;68(8):1231-1253. doi: 10.1007/s12630-021-02015-0. Epub 2021 May 19. PMID 34013463
- [Background] Padmanabhan R, Hildreth AJ, Laws D. A prospective, randomised, controlled study examining binaural beat audio and pre-operative anxiety in patients undergoing general anaesthesia for day case surgery. Anaesthesia. 2005 Sep;60(9):874-7. doi: 10.1111/j.1365-2044.2005.04287.x. PMID 16115248
- [Background] Wiwatwongwana D, Vichitvejpaisal P, Thaikruea L, Klaphajone J, Tantong A, Wiwatwongwana A; Medscape. The effect of music with and without binaural beat audio on operative anxiety in patients undergoing cataract surgery: a randomized controlled trial. Eye (Lond). 2016 Nov;30(11):1407-1414. doi: 10.1038/eye.2016.160. Epub 2016 Oct 14. PMID 27740618
- [Background] Bae J, Yoo S, Kim H, Kim Y, Kim JT, Lim YJ, Kim HS. Effect of real-time binaural music on sedation with dexmedetomidine during spinal anesthesia: A triple-arm, assessor-blind, randomized controlled trial. J Clin Anesth. 2023 Feb;84:110997. doi: 10.1016/j.jclinane.2022.110997. Epub 2022 Nov 10. PMID 36371942
- [Background] Schmid W, Marhofer P, Opfermann P, Zadrazil M, Kimberger O, Triffterer L, Marhofer D, Klug W. Brainwave entrainment to minimise sedative drug doses in paediatric surgery: a randomised controlled trial. Br J Anaesth. 2020 Sep;125(3):330-335. doi: 10.1016/j.bja.2020.05.050. Epub 2020 Jul 8. PMID 32653082
- [Background] Facco E, Stellini E, Bacci C, Manani G, Pavan C, Cavallin F, Zanette G. Validation of visual analogue scale for anxiety (VAS-A) in preanesthesia evaluation. Minerva Anestesiol. 2013 Dec;79(12):1389-95. Epub 2013 Jul 9. PMID 23860442
- [Background] Long MHY, Lim EHL, Balanza GA, Allen JC Jr, Purdon PL, Bong CL. Sevoflurane requirements during electroencephalogram (EEG)-guided vs standard anesthesia Care in Children: A randomized controlled trial. J Clin Anesth. 2022 Oct;81:110913. doi: 10.1016/j.jclinane.2022.110913. Epub 2022 Jun 27. PMID 35772250